CLINICAL TRIAL: NCT02555605
Title: Feasibility of Dexmedetomidine in Children With Respiratory Morbidities Undergoing Deep Sedation for Magnetic Resonance Imaging
Brief Title: Dexmedetomidine Sedation in Children With Respiratory Morbidities
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Other Study IDs: DEXMRI20
Record Dates: First submitted 2015-08-11; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Respiratory Morbidity
Keywords: children; dexmedetomidine; magnetic resonance imaging scans; deep sedation; adverse respiratory events
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexmedetomidine — Children up to the age of 16 years requiring MRI under deep sedation with at least 3 characteristics of respiratory morbidities were identified as having increased risk for adverse respiratory events. Dexmedetomidine was administered as a first bolus of 1 mcg•kg-1 over 10 min, followed by a continuous infusion at 1.0 mcg•kg-1•h-1. Sedation level was assessed by Ramsay Sedation Scale and it was initially recorded at 1-min interval. If the child failed to achieve a minimum RSS of 5, this bolus was repeated once again and the continuous infusion was subsequently increased to 2 mcg•kg-1•h-1. In addition, propofol 0.5 mg.kg-1 iv. was allowed to be administered, in patients still exhibiting movement that could interfere with image acquisition.
  Other Names: Dexdor

SUMMARY:
This study aimed to determine the feasibility of dexmedetomidine in children with respiratory morbidities who required deep sedation for magnetic resonance imaging (MRI) scans.

DETAILED DESCRIPTION:
Electronic medical records of children with at least 3 characteristics of respiratory morbidities were retrospectively reviewed. All study patients received dexmedetomidine bolus over 10 min followed by a continuous infusion to achieve a minimum Ramsay Sedation Score of 5. Patients were monitored for hemodynamics, total dose of dexmedetomidine received, adverse events experienced and sedation characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Children up to the age of 16 years with at least 3 characteristics of respiratory morbidities

Exclusion Criteria:

* Children who had an American Society of Anaesthesiologists (ASA) physical status classification IV
* Documented pre-existing cardiac conduction abnormalities
* Renal impairment

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children up to the age of 16 years with at least 3 characteristics of respiratory morbidities were identified as having increased risk for adverse respiratory events and they were eligible for participation in this evaluation.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the occurrence of successful sedation | 1 hour
  completion of imaging without requirement for rescheduling or general anaesthesia, and in the absence of adverse respiratory events such as apnoea, cough, oxygen desaturation, and bronchospasm or unplanned escalation of care (e.g. transfer from ward to paediatric intensive care unit or prolonged hospitalization).

SECONDARY OUTCOMES:
the presence of bradycardia | 4 hours
  Based on age-adjusted criteria, bradycardia was defined as a HR <20% below the lower limit of the normal ranges expressed in beats/min
the presence of hypertension | 4 hours
  Based on age-adjusted criteria hypertension was defined as a MAP >20% above the upper limit of the normal ranges expressed in mmHg
the presence of nausea and vomiting. | 4 hours
  defined as the occurrence of nausea and vomitting, expressed in "yes" or "no"

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Najafi, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Jan Poelaert, PhD MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Najafi N, Veyckemans F, Van de Velde A, Poelaert J. Usability of dexmedetomidine for deep sedation in infants and small children with respiratory morbidities. Acta Anaesthesiol Scand. 2016 Aug;60(7):865-73. doi: 10.1111/aas.12715. Epub 2016 Mar 4. PMID 26940080